CLINICAL TRIAL: NCT06263049
Title: Ejaculatory Preserving Transurethral Resection of the Prostate.
Brief Title: Is Ejaculation Preservation TURis the Natural Evolution of the "Gold Standard".
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ejaculation post TURP
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: ejaculation, incontinence
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): (TURP group underwent traditional TURP)
  Interventions: Procedure: transurethral resection of prostate
- group B (Active Comparator): TURP with preserved urethral mucosa at the prostatic apex
  Interventions: Procedure: transurethral resection of prostate

INTERVENTIONS:
Procedure: transurethral resection of prostate — resection of prostate by using bipolar cautarization

SUMMARY:
evaluation of the impact of apical urethral mucosa sparring with the urethra around the verumontanum on the ejaculatory function and early postoperative urinary incontinence

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) is a common disease in elderly men and transurethral resection of the prostate (TURP) is still the gold standard for the treatment of BPH However, postoperative urinary incontinence (UI) and retrograde ejaculation are of the common complications and its incidence is nearly 2% of UI UI brings great suffering to patients and its unpredictability and uncertainty in the recovery period cause significant pressure to surgeons. External urethral sphincter damage is the main reason for UI after prostatectomy. The treatment of postoperative UI and post operative retrograde ejaculation has also become an important issue for many years. Along with the progress of technology, there have been various methods of transurethral resection of the prostate but no method has been found to adequately avoid the occurrence of UI and retrograde ejaculation

ELIGIBILITY:
Our inclusion criteria were preidentified to those who complained of voiding lower urinary tract symptoms (LUTS) and scheduled for TURP with prostate size less than 100 gm. This included patients with refractory retention, recurrent gross hematuria of prostatic origin, non-compliance to medical treatment, recurrent infection, and patients with bladder calculi secondary to obstruction. Exclusion criteria were: patients with neurogenic bladder, detrusor hypo-contractility, Diabetes more than 10 years, urethral stricture, or previous prostatic surgeries.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
post operative antegrade ejaculation | within 1 month post operative
  the ability of the person to ejaculate post TURP procedure

SECONDARY OUTCOMES:
post operative urine continence | within 1 month post operative
  early postoperative urine continence

CONTACTS AND LOCATIONS:
Overall Officials: mohamed essmat aboughareb, consultant, Study Director — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liang JQ, Ma WT, Lu BW, Dai L, Zhao YM, Zhang JD, Tian B, Liu QL. Clinical Study on the Application of Preserved Urethral Mucosa at the Prostatic Apex in Transurethral Plasmakinetic Resection of the Prostate. Front Surg. 2022 Jun 17;9:922479. doi: 10.3389/fsurg.2022.922479. eCollection 2022. PMID 35784938